CLINICAL TRIAL: NCT01011257
Title: Methods to Augment the Efficacy of Aspirin and Clopidogrel in Healthy Subjects (ASA Only) and Patients With Stable Coronary Artery Disease (Taking Clopidogrel Only) or (Taking Clopidogrel & ASA) With an Elevated Platelet Turnover (Reticulated Platelets).
Brief Title: Studying the Efficacy of Aspirin & Clopidogrel in Healthy Subjects With Stable Coronary Artery Disease.
Acronym: Dual-Dosing
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding secured.
Sponsor: Neil Kleiman, MD (Other)
Responsible Party: Sponsor-Investigator, Neil Kleiman, MD, Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001863
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — acetylsalicylic acid lysinate; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin 81 mg, 1 tab twice daily (Active Comparator): All participants to take one aspirin (81mg per tab) twice daily.
  Interventions: Drug: Asprin
- Clopidogrel 75 mg 1 tab daily (Active Comparator): Only stable CAD participants will take Clopidogrel (75mg per tab) daily.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Asprin — asprin 81mg, 1 tab, twice daily OR aspirin 81mg, 2 tab, once daily
  Other Names: ASA
  Arms: Aspirin 81 mg, 1 tab twice daily
Drug: Clopidogrel — clopidogrel 75 mg bid
  Other Names: Plavix
  Arms: Clopidogrel 75 mg 1 tab daily

SUMMARY:
The investigators will test the hypothesis that aspirin or clopidogrel taken twice daily will augment their antiplatelet efficacy in patients with an elevated platelet turnover (as measured by the proportion of reticulated (young) platelets) compared with once daily dosing.

DETAILED DESCRIPTION:
1. To study whether in healthy subjects with an increased platelet turnover, a twice daily dosing of aspirin 81 mg will be more effective in inhibiting platelets compared with once a day aspirin 81 mg.
2. To study whether in patients with stable coronary artery disease (CAD) with an increased platelet turnover, a twice daily dosing of aspirin 81 mg will be more effective in inhibiting platelets compared with once a day aspirin 81 mg.
3. To study whether in healthy subjects with an increased platelet turnover, a twice daily dosing of aspirin 81 mg and clopidogrel 75 mg will be more effective in inhibiting platelets compared with once daily of both aspirin and clopidogrel.
4. To study whether in patients with stable coronary artery disease (CAD), increased platelet turnover and aspirin resistance, an oral fatty acid (docosahexaenoic acid (DHA) and eicosapentanoic acid (EPA), 4 gm/day) supplementation will increase the efficacy of aspirin by modifying platelet function compared to once a day aspirin 81 mg.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Healthy subjects aged 18-64 years with no evidence of coronary artery disease or any major risk factors for CAD including smoking, diabetes mellitus, hyperlipidemia, hypertension and obesity.
* Group B: Patients with known CAD aged 18-64 years taking aspirin 81 mg daily as the only antiplatelet therapy. Patients should be in stable condition and at least one month post myocardial infarction.
* Group C: Patients with known stable CAD aged 18-64 years taking aspirin 81 mg and clopidogrel 75 mg daily. Patients should be in stable condition and at least one month post myocardial infarction.

Exclusion Criteria:

* Subjects will be excluded if they used NSAID's within one week prior to the study, have renal insufficiency, inflammatory disorders such as rheumatologic conditions, autoimmune disorders, active infections, malignancy or if they are undergoing chemotherapy.
* Other exclusion criteria include contraindications to aspirin including active bleeding, hypersensitivity, thrombocytopenia (platelet count < 50,000) and anemia (hemoglobin < 10.0 gm/dl).
* We will also exclude patients with unstable angina and recent (less than a month) CABG or PCTA.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To look if dual dosing of aspirin and/or clopidogrel will augment antiplatelet efficacy in patients with elevated reticulated platelet turnover. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Kleiman, MD, Principal Investigator — Methodist DeBakey Heart Center.
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No